CLINICAL TRIAL: NCT01580228
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Dinaciclib or Ofatumumab in Subjects With Refractory Chronic Lymphocytic Leukemia
Brief Title: A Phase 3 Study Comparing Dinaciclib Versus Ofatumumab in Patients With Refractory Chronic Lymphocytic Leukemia (P07714)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P07714; 2011-005186-20 (EudraCT Number)
Record Dates: First submitted 2012-04-03; First posted 2012-04-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — dinaciclib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dinaciclib (Experimental)
  Interventions: Drug: Dinaciclib
- Ofatumumab (Active Comparator)
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Dinaciclib — Dinaciclib administered intravenously over 2 hours at a dose of 7 mg/m^2 on Day 1, 10 mg/m^2 on Day 8, and 14 mg/m^2 on Day 15 in Cycle 1. Starting in Cycle 2 and thereafter, dinaciclib will be dosed at 14 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle for a total of 12 cycles.
  Other Names: SCH-727965; MK-7965
  Arms: Dinaciclib
Drug: Ofatumumab — Ofatumumab administered intravenously at a dose of 300 mg on Cycle 1 Day 1, followed by 2000 mg on Cycle 1 Days 8, 15, and 22; Cycle 2 Days 1, 8, 15, and 22; followed 5 weeks later on Day 1 of Cycles 4-12.
  Other Names: Arzerra
  Arms: Ofatumumab

SUMMARY:
This study is being conducted to demonstrate the superiority in progression-free survival (PFS) of dinaciclib compared to ofatumumab in chronic lymphocytic leukemia (CLL) participants with del 17p or in the overall population who are refractory to either fludarabine treatment or chemoimmunotherapy.

DETAILED DESCRIPTION:
Dinaciclib is a cyclin-dependent kinase (CDK) inhibitor, specific for CDK 1, 2, 5 and 9.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL)
* Fludarabine or chemoimmunotherapy refractory disease defined as: failing to respond to or relapsed within 6 months of completing fludarabine or another purine analog alone or in combination regimens, or failing to respond to chemoimmunotherapy or relapsed within 24 months of completing therapy with a combination of chemotherapy plus an anti-CD20 monoclonal antibody
* Eastern Cooperative Oncology Group (ECOG) Performance status 0, 1, or 2
* Adequate organ function and laboratory parameters
* Women of child-bearing potential who are not currently sexually active must

agree to use a medically accepted method of contraception should they become

sexually active while participating in the study

Exclusion Criteria:

* Symptomatic brain metastases or primary central nervous system malignancy
* Treatment with a CYP3A4 inhibitor or inducer within 1 week prior to randomization, or any chemotherapy or biologic therapy within 4 weeks prior to randomization
* Known human immunodeficiency virus (HIV) infection or a known HIV-related

malignancy

* Participants with with clinically active hepatitis B or C defined as disease that requires therapy
* Positive test for glucose-6 phosphate dehydrogenase (G6PD) deficiency
* Prior allogeneic bone marrow transplant
* Presence of Richter's transformation
* Indeterminate deletion 17p status
* Previous treatment with ofatumumab, dinaciclib, or other CDK inhibitors
* Active autoimmune anemia or thrombocytopenia unless stable, which is defined as being responsive to corticosteroids or other standard therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Participant Progression Free Survival | From date of randomization up to approximately 38 months

SECONDARY OUTCOMES:
Participant Overall Response Rate | From date of randomization up to approximately 38 months
Participant Overall Survival Rate | From date of randomization until up to approximately 50 months

REFERENCES:
- [Result] Ghia P, Scarfo L, Perez S, Pathiraja K, Derosier M, Small K, McCrary Sisk C, Patton N. Efficacy and safety of dinaciclib vs ofatumumab in patients with relapsed/refractory chronic lymphocytic leukemia. Blood. 2017 Mar 30;129(13):1876-1878. doi: 10.1182/blood-2016-10-748210. Epub 2017 Jan 26. No abstract available. PMID 28126927